CLINICAL TRIAL: NCT00227149
Title: Long-Term Evaluation Follow-up of Neurocognitive Performance and Emotional State in Patients With Chronic Hepatitis C Infection and a Former (Peg)Interferon Alfa-2b-Based Therapy
Brief Title: Long-Term Evaluation Follow-up of Neurocognitive Performance and Emotional State in Patients With Chronic Hepatitis C
Status: Completed | Type: Observational
Sponsor: University of Wuerzburg (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Michael R Kraus, MD, PhD, University of Wuerzburg
Other Study IDs: PO 4406
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Hepatitis C, Chronic
Keywords: C06.552.380.705.440
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a long-term evaluation follow-up study of neurocognitive performance and emotional state in patients with chronic hepatitis C infection and a former (peg)interferon alfa-2b-based therapy.

M.R. Kraus, G. Teuber, NN, NN (MPsych), M. Scheurlen

Questions:

* Neurocognitive and psychiatric changes induced by interferon alfa-2b therapy in patients with chronic hepatitis C - are they fully reversible in long-term follow-up after the end of antiviral treatment?
* At least 12 months after the end of antiviral treatment - are neurocognitive and mood-related parameters even significantly improved as compared to pretreatment values? Is this possibly only true of patients with successful virus eradication?
* At least 12 months after the end of antiviral treatment, is there a significant difference between patients with and without sustained virological response with respect to neurocognitive performance, emotional state and quality of life?
* In the absence of clinically significant liver damage in patients with chronic hepatitis C - does the mere presence of the hepatitis C virus have any significant influence on neurocognitive or attentional performance?
* Does the study data support an additional indication for antiviral therapy in chronic hepatitis C? In the case of successful virus eradication, emotional state and - above all - is neurocognitive performance significantly improved even in the absence of severe liver damage?

DETAILED DESCRIPTION:
This is a long-term evaluation follow-up study of neurocognitive performance and emotional state in patients with chronic hepatitis C infection and a former (peg)interferon alfa-2b-based therapy.

M.R. Kraus, G. Teuber, NN, NN (MPsych), M. Scheurlen

Questions:

* Neurocognitive and psychiatric changes induced by interferon alfa-2b therapy in patients with chronic hepatitis C - are they fully reversible in long-term follow-up after the end of antiviral treatment?
* At least 12 months after the end of antiviral treatment - are neurocognitive and mood-related parameters even significantly improved as compared to pretreatment values? Is this possibly only true of patients with successful virus eradication?
* At least 12 months after the end of antiviral treatment, is there a significant difference between patients with and without sustained virological response with respect to neurocognitive performance, emotional state and quality of life?
* Can the results of the current and previous studies be confirmed by alternative / additional psychometric instruments in specified subsample? (Fatigue Impact Scale; FIS-D, SF-36)
* In the absence of clinically significant liver damage in patients with chronic hepatitis C - does the mere presence of the hepatitis C virus have any significant influence on neurocognitive or attentional performance?
* Does the study data support an additional indication for antiviral therapy in chronic hepatitis C? In the case of successful virus eradication, is emotional state and - above all - neurocognitive performance significantly improved even in the absence of severe liver damage?

Methods:

* Multifactorial analysis of test results: pre- vs. post-therapy; sustained virological response vs. nonresponse/relapse.
* Psychometric evaluation instruments / psychometric questionnaires (HADS-D, SCL-90-R, Subsample : SF-36, FIS-D)
* Evaluation of neurocognitive performance by the Test battery of Attentional Performance (TAP)
* Evaluation in a prospective, longitudinal study design.

Planned sample size / sample size considerations

* N = 150 patients (hepatitis C patients in a longitudinal study design: t1[before onset of interferon therapy] … t5[at least 12 months after the end of antiviral treatment]

Power calculations / power considerations:

* Given: 2-factorial design (time course x SVR); type I error = 0.050; type II error = 0.20 (power = 0.80) - as usually assumed in clinical trials.
* With respect to the independent factor SVR ("sustained virological response", 2 factor levels), optimum / optimal sample sizes range from 42 (large effect size d = 0.8) to 102 (medium effect size d = 0.5). Smaller effect sizes - according to previous work in this field - do not appear to bear any clinical relevance.
* (Pairwise comparisons of dependent samples [e.g. pre- vs. post-therapy or pre-therapy vs. long-term follow-up] require even smaller optimal sample sizes ranging from 16 to 43 for large or medium effect sizes.)

Patient recruitment:

* Patients with chronic hepatitis C infection and therapy with (peg)interferon alfa-2b.
* Patients with informed written consent (with respect) to a long-term follow-up of psychiatric side effects and neurocognitive performance.
* Patients with baseline monitoring of neuropsychiatric symptoms and neurocognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis C and indication for interferon-based antiviral therapy.
* Written informed consent to study participation, especially to long-term follow-up monitoring of psychiatric and neurocognitive side effects of combination therapy with (peg)interferon alfa-2b and ribavirin.
* Age of study participants: between 18 and 65 years.
* All patients need to have documented antibodies to hepatitis C virus (HCV) and circulating HCV-RNA as measured by reverse-transcription polymerase chain reaction (Cobas Amplicor HCV Monitor™ test, Roche Diagnostics)

Exclusion Criteria:

* Insufficient knowledge of the German language or cognitive impairment (due to the indispensable application of questionnaires and the TAP, test battery of attentional performance).

Further Exclusion Criteria:

* Age under 18 years or over 65 years
* Coinfections such as hepatitis B virus or human immunodeficiency virus
* Severe internal diseases (e.g., cancer, ischemic heart disease, autoimmune disease)
* Major depressive disorder (according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition [DSM-IV] criteria), psychosis, active intravenous drug use or alcohol abuse.

These additional exclusion criteria are important in order to avoid interfering or confounding effects by other variables that are not linked to the hepatitis C infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCV outpatients (University Hospital)
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2005-07; Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Kraus, MD, PhD, Principal Investigator — Med. Klinik und Poliklinik II, University of Wuerzburg
Locations (1):
- Med. Klinik und Poliklinik II, University of Wuerzburg, Würzburg, Germany

REFERENCES:
- [Background] Kraus MR, Schafer A, Wissmann S, Reimer P, Scheurlen M. Neurocognitive changes in patients with hepatitis C receiving interferon alfa-2b and ribavirin. Clin Pharmacol Ther. 2005 Jan;77(1):90-100. doi: 10.1016/j.clpt.2004.09.007. PMID 15637534
- [Background] Kraus MR, Schafer A, Faller H, Csef H, Scheurlen M. Psychiatric symptoms in patients with chronic hepatitis C receiving interferon alfa-2b therapy. J Clin Psychiatry. 2003 Jun;64(6):708-14. doi: 10.4088/jcp.v64n0614. PMID 12823087
- [Background] Kraus MR, Schafer A, Faller H, Csef H, Scheurlen M. Paroxetine for the treatment of interferon-alpha-induced depression in chronic hepatitis C. Aliment Pharmacol Ther. 2002 Jun;16(6):1091-9. doi: 10.1046/j.1365-2036.2002.01265.x. PMID 12030950
- [Background] Kraus MR, Schafer A, Scheurlen M. Paroxetine for the prevention of depression induced by interferon alfa. N Engl J Med. 2001 Aug 2;345(5):375-6. No abstract available. PMID 11484704